CLINICAL TRIAL: NCT03214822
Title: The Impact of Human-derived Human Milk Fortifiers (H2MF) on Gut Microbiota Development and Oxidative Stress in Premature Infants
Brief Title: Human-derived Human Milk Fortifiers (H2MF), Gut Microbiota and Oxidative Stress in Premature Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Manitoba Developmental Origins of Chronic Diseases in Children Network (DEVOTION) (Unknown); Prolacta Bioscience (Industry); Children's Hospital Foundation (Other)
Responsible Party: Principal Investigator, Meghan Azad, Prinicpal Investigator, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: H2MF Study
Record Dates: First submitted 2017-07-05; First posted 2017-07-12 (Actual); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Very Low Birth Weight Baby; Premature Birth; Microbial Colonization; Oxidative Stress
Keywords: Microbiome
MeSH Terms: conditions — Premature Birth; Communicable Diseases

STUDY DESIGN:
Intervention Model Description: Using a randomized, controlled, un-blinded parallel design we will enroll 30 VLBW premature neonates (birth weight < 1250 grams, gestational age 26+0 to 30+0 weeks) from the NICU at the Health Sciences Centre Children's Hospital in Winnipeg, MB, Canada. Currently, H2MF is not routinely used in this population at this centre.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Masking of care providers is not feasible since the procedures of preparation for HMF and H2MF are different. Outcome assessors (personnel analyzing microbiome profiles and oxidative stress biomarkers) will be masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- HMF (standard of care) (No Intervention): The HMF "Control Group" will receive the current standard feeding protocol of human milk fortified with bovine (cow) human milk fortifier (HMF)
- H2MF (Experimental): The H2MF "Intervention Group" will receive identical treatment with human-derived human milk fortifier (H2MF) replacing standard bovine HMF until the baby reaches an adjusted gestation age of 33 weeks; followed by a 5 day ween to standard HMF according to the manufacturer's recommendation.
  Interventions: Dietary Supplement: H2MF

INTERVENTIONS:
Dietary Supplement: H2MF — As described in the Experimental Arm description.
  Arms: H2MF

SUMMARY:
This is a randomized controlled trial of a human-derived human milk fortifier (H2MF) vs standard bovine-derived human milk fortifier (HMF) evaluating fecal microbiota and fecal and urinary biomarkers of oxidative stress in premature infants.

DETAILED DESCRIPTION:
While breast milk provides complete nutrition for full term infants, supplementation with human milk fortifiers (HMF) is required to achieve optimal weight gain in very low birthweight (VLBW) preterm neonates. Traditionally, HMF have been derived from bovine milk. Bovine-based infant formula has been shown to cause dysbiosis of the infant gut microbiome (Azad et al 2013) and increased oxidative stress in preterm neonates (Friel et al 2011). Microbiome dysbiosis and oxidative stress have been implicated in numerous inflammatory conditions, including both acute (eg. necrotizing enterocolitis, NEC) and long-term (eg. asthma, metabolic syndrome) sequela of preterm birth (Torrazza et al 2013, Goulet et al 2015, Flora et al 2007, Perrone et al 2014). Recent studies show that new human-derived HMF (H2MF) are superior to standard bovine HMF for nourishing VLBW preterm infants and preventing NEC (Sullivan et al 2010, Cristofalo et al 2013). However, the biological basis for these clinical benefits is unknown, which limits our ability to inform and improve feeding strategies for VLBW preterm infants. This will be the first study to evaluate the impact of H2MF on gut microbiota and oxidative stress in preterm infants.

Specific Objectives:

1. To evaluate the effect of H2MF vs. HMF on gut microbiota composition in premature infants born <1250 gr between 26 and 30 weeks of gestational age.
2. To evaluate the effect of H2MF vs. HMF on fecal and urinary biomarkers of oxidative stress in premature infants born <1250 gr between 26 and 30 weeks of gestational age.

ELIGIBILITY:
Inclusion Criteria:

* Male or female infant with birth weight <1250 grams
* Gestational age between 26+0 to 30+0 weeks at birth
* Able to adhere to feeding protocol
* Parenteral nutrition must be started by day of life 2
* Enteral feeding >80 ml/kg/d should be reached by day of life 14
* Subject's parent(s)/legal guardian(s) has provided signed and dated informed consent and authorization to use protected health information, as required by national and local regulations.
* In the investigator's opinion, the subject's parent(s)/legal guardian(s) understands and is able to comply with protocol requirements, instructions, and protocol-stated restrictions, and is likely to complete the study as planned.

Exclusion Criteria:

* Gestational age > 30+0 weeks at birth (to guarantee a minimum of 3 weeks H2MF treatment, since fortification ends at 33+0 AGA)
* Gestational age < 26+0 weeks at birth (to minimize baseline heterogeneity, since gestational age influences gut microbiota)
* Received antibiotics on the first day of specimen collection (to minimize baseline heterogeneity, since antibiotics influence gut microbiota) Note: all infants are expected to receive up to 48 hr antibiotic prophylaxis at birth according to standard NICU protocol; this criterion will exclude infants receiving extended courses of antibiotics.
* Received probiotics at any time (to minimize baseline heterogeneity, since probiotics influence gut microbiota)
* Unlikely to survive the study period
* Presence of clinically significant congenital heart disease or other major congenital malformation
* Presence prior to enrollment of intestinal perforation or stage 2 necrotizing enterocolitis (NEC) prior to tolerating fortified feeds

Max Age: 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
Fecal microbiome composition at end of intervention | 33+0 weeks adjusted gestational age (end of intervention)
  Relative abundance of operational taxonomic units (OTUs) determined by 16S rRNA Illumina sequencing
Fecal microbiome diversity at end of intervention | 33+0 weeks adjusted gestational age (end of intervention)
  Shannon diversity index of microbiota, determined by 16S rRNA Illumina sequencing
Fecal microbiome community structure at end of intervention | 33+0 weeks adjusted gestational age (end of intervention)
  Principal coordinate analysis using UniFrac distance matrices based on 16S rRNA Illumina sequencing

SECONDARY OUTCOMES:
Fecal microbiome at 1 week after intervention begins | Study day 7 (1 week after intervention begins)
  Fecal microbiome composition, diversity and community structure from 16S rRNA Illumina Sequencing.
Fecal microbiome at 2 weeks after intervention ends | 35+0 weeks adjusted gestational age (2 weeks after intervention ends)
  Fecal microbiome composition, diversity and community structure from 16S rRNA Illumina Sequencing.
Oxidative stress (urinary biomarkers) at end of intervention | 33+0 weeks adjusted gestational age (end of intervention)
  F2-isoprostanes, 8-hydroxy deoxyguanine, and visfatin measured in urine.
Oxidative stress (fecal calprotectin) at end of intervention | 33+0 weeks adjusted gestational age (end of intervention)
  Calprotectin measured in feces
Oxidative stress at 1 week after intervention begins | Study day 7 (1 week after intervention begins)
  Fecal and urinary biomarkers of oxidative stress (fecal calprotectin, urinary F2-isoprostanes, urinary 8-hydroxy deoxyguanine, urinary visfatin).
Oxidative stress at 2 weeks after intervention ends | 35+0 weeks adjusted gestational age (2 weeks after intervention ends)
  Fecal and urinary biomarkers of oxidative stress (fecal calprotectin, urinary F2-isoprostanes, urinary 8-hydroxy deoxyguanine, urinary visfatin).

CONTACTS AND LOCATIONS:
Overall Officials: Meghan Azad, PhD, Principal Investigator — University of Manitoba; Geert T'Jong, Study Director — University of Manitoba
Locations (1):
- Health Sciences Centre, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: Undecided
At this time we plan to share IPD within our research team only. We will consider sharing with other researchers in the future.

REFERENCES:
- [Background] Azad MB, Konya T, Maughan H, Guttman DS, Field CJ, Chari RS, Sears MR, Becker AB, Scott JA, Kozyrskyj AL; CHILD Study Investigators. Gut microbiota of healthy Canadian infants: profiles by mode of delivery and infant diet at 4 months. CMAJ. 2013 Mar 19;185(5):385-94. doi: 10.1503/cmaj.121189. Epub 2013 Feb 11. PMID 23401405
- [Background] Friel JK, Diehl-Jones B, Cockell KA, Chiu A, Rabanni R, Davies SS, Roberts LJ 2nd. Evidence of oxidative stress in relation to feeding type during early life in premature infants. Pediatr Res. 2011 Feb;69(2):160-4. doi: 10.1203/PDR.0b013e3182042a07. PMID 21045751
- [Background] Torrazza RM, Ukhanova M, Wang X, Sharma R, Hudak ML, Neu J, Mai V. Intestinal microbial ecology and environmental factors affecting necrotizing enterocolitis. PLoS One. 2013 Dec 30;8(12):e83304. doi: 10.1371/journal.pone.0083304. eCollection 2013. PMID 24386174
- [Background] Goulet O. Potential role of the intestinal microbiota in programming health and disease. Nutr Rev. 2015 Aug;73 Suppl 1:32-40. doi: 10.1093/nutrit/nuv039. PMID 26175488
- [Background] Flora SJ. Role of free radicals and antioxidants in health and disease. Cell Mol Biol (Noisy-le-grand). 2007 Apr 15;53(1):1-2. No abstract available. PMID 17535753
- [Background] Perrone S, Tataranno ML, Santacroce A, Negro S, Buonocore G. The role of oxidative stress on necrotizing enterocolitis in very low birth weight infants. Curr Pediatr Rev. 2014;10(3):202-7. PMID 25088341
- [Background] Sullivan S, Schanler RJ, Kim JH, Patel AL, Trawoger R, Kiechl-Kohlendorfer U, Chan GM, Blanco CL, Abrams S, Cotten CM, Laroia N, Ehrenkranz RA, Dudell G, Cristofalo EA, Meier P, Lee ML, Rechtman DJ, Lucas A. An exclusively human milk-based diet is associated with a lower rate of necrotizing enterocolitis than a diet of human milk and bovine milk-based products. J Pediatr. 2010 Apr;156(4):562-7.e1. doi: 10.1016/j.jpeds.2009.10.040. Epub 2009 Dec 29. PMID 20036378
- [Background] Cristofalo EA, Schanler RJ, Blanco CL, Sullivan S, Trawoeger R, Kiechl-Kohlendorfer U, Dudell G, Rechtman DJ, Lee ML, Lucas A, Abrams S. Randomized trial of exclusive human milk versus preterm formula diets in extremely premature infants. J Pediatr. 2013 Dec;163(6):1592-1595.e1. doi: 10.1016/j.jpeds.2013.07.011. Epub 2013 Aug 20. PMID 23968744
- [Derived] Kumbhare SV, Jones WD, Fast S, Bonner C, Jong G', Van Domselaar G, Graham M, Narvey M, Azad MB. Source of human milk (mother or donor) is more important than fortifier type (human or bovine) in shaping the preterm infant microbiome. Cell Rep Med. 2022 Sep 20;3(9):100712. doi: 10.1016/j.xcrm.2022.100712. Epub 2022 Aug 26. PMID 36029771